CLINICAL TRIAL: NCT02512458
Title: A Study of Cabazitaxel Treatment in Castration Resistant Bone Metastatic Prostate Cancer Patients Evaluating the Tumor Microenvironment
Brief Title: Study of the Effect of Chemotherapy With Cabazitaxel on Prostate Cancer
Acronym: CABA-BONE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE 9A/14; 2014-004485-21 (EudraCT Number)
Record Dates: First submitted 2015-07-21; First posted 2015-07-31 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Bone Metastatic Prostate Cancer
MeSH Terms: interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel (Experimental): Patient will be treated with iv cabazitaxel 25mg/m2 q 21days per standard clinical practice for up to 10 cycles or until disease progression or unacceptable toxicity or physician's decision or patient's consent withdrawal (whichever occurs first).
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel
  Other Names: Jevtana

SUMMARY:
This is a prospective, open-label, single arm translational study of cabazitaxel in bone Castration Resistant metastatic Pancreatic Cancer (mCRPC) patients. Patient will be treated with intravenous (iv) cabazitaxel 25mg/m2 every (q) 21days per standard clinical practice for up to 10 cycles or until disease progression or unacceptable toxicity or physician's decision or patient's consent withdrawal (whichever occurs first).

DETAILED DESCRIPTION:
This is an open-label, interventional study to explore the effect of Cabazitaxel on survival pathways and androgen signaling in the tumor microenvironment (bone marrow) of patients with castration resistant metastatic prostate cancer.

A total of 30 evaluable patients are needed. An estimated 50% chance of failure to harvest evaluable bone marrow biopsy or aspirate is anticipated based on investigators prior experience. Thus a total of 60 patients will be accrued in the study. This will provide the investigators an 80% power to detect an effect size of at least 0.82, using a two-sided paired t-test and at a 0.05 significance level.The changes in androgen signaling (androgen receptor expression and other survival pathway markers, between baseline and 9 weeks will be assessed by paired t-test and Wilcoxon signed-rank test. The association between serum Prostate-Specific Androgen (PSA) and bone marrow androgen signaling level will be evaluated using scatter plot and spearman's correlation coefficient. Similar methods will be used to explore the association between circulating androgens and those in the bone marrow.

Biomarker data will also be summarized and compared between baseline and after treatment using paired t-test or Wilcoxon signed-rank test.

ECOG changes from baseline will be provided for each treatment period. All Adverse Events (AE) will be graded using the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) classification, version 4.3.

Summary tables of Adverse Events (AE)s, Treatment Emergent Adverse Event(TEAE), Serious Adverse Events (SAE)s and withdrawals for adverse events will be provided by treatment period. Adverse events will be summarized by worst severity grade AEs.

All registered subjects who take at least 1 dose of agent will be included in the safety analyses. Adverse events will be summarized by worst severity grade. AEs, as well as treatment-emergent AEs, will be summarized by system organ class, and preferred term. Investigational Medicinal Products (IMP) -related adverse events, adverse events leading to death or to discontinuation from treatment, events classified as NCI-CTCAE v4 Grade 3 or Grade 4 (or moderate/severe if other rating scale is used), (IMP)-related events, and serious adverse events will be summarized separately.

ELIGIBILITY:
Inclusion Criteria:

* Male patients older than 18 years
* Histologically proven adenocarcinoma of the prostate
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Serum testosterone levels < 50ng/ml (1.7 nmol/L)
* Ongoing gonadal androgen deprivation therapy with Luteinizing Hormone-Releasing Hormone (LHRH) analogues or orchiectomy. Patients, who have not had an orchiectomy, must be maintained on effective LHRH analogue therapy for the duration of the trial
* Progression of disease despite androgen ablation - Either documented osseous or soft tissue metastatic disease progression or by PSA criteria progression
* Presence of bone metastases
* Off diethylstilbestrol (DES) or steroids treatment for ≥ 4 weeks and for antiandrogens > 4 weeks.
* No prior treatment with cabazitaxel
* Able to comply with study requirements
* Written information delivered to the patient. Patient must be willing and able to comply with protocol requirements. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must also have signed an authorization for the release of their protected health information.

Exclusion Criteria:

* Histologic variants in the primary tumor (histologic variants other than adenocarcinoma)
* Concurrent therapy with other therapeutic or hormonal agent, including androgen receptor antagonists (bicalutamide, flutamide, nilutamide, enzalutamide), any dose of megestrol acetate (Megace), ketoconazole, abiraterone acetate, finasteride (Proscar), dutasteride (Avodart) any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES),
* Active infection or intercurrent illnesses that are not controlled
* Prior radiation therapy completed < 4 weeks prior to enrolment
* Planned palliative procedures for alleviation of bone pain such as radiation therapy or surgery
* Structurally unstable bone lesions suggesting impending fracture
* Any "currently active" second malignancy, other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy, if they have completed therapy and are considered by their physician to be at least less than 30% risk of relapse over next 3 months
* Active psychiatric illnesses/social situations that would limit compliance with protocol requirements.
* Active or uncontrolled autoimmune disease that may require corticosteroid therapy during study.
* Severely compromised immunological state, including being positive for the human immunodeficiency virus (HIV)
* Known acute or chronic hepatitis B or C
* Other investigational therapies (targeted or vaccine) will require a 4 week washout period before treatment initiation
* Ιnitiation of bisphosphonate or denosumab therapy within 4 weeks prior to first dose of study drug. Patients on stable doses of bisphosphonates or denosumab that show subsequent tumor progression may continue on this medication; however, patients are discouraged to initiate bisphosphonate therapy during the study.
* Patients receiving an investigational drug within 4 weeks prior to enrolment
* History of severe hypersensitivity reaction (grade ≥3) to polysorbate 80 containing drugs
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus)
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments)
* Inadequate organ or bone marrow function

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Molecular effects of treatment with Cabazitaxel on the tumor microenvironment | On week 9 and on week 36
  To explore molecular effects of treatment with Cabazitaxel on the tumor microenvironment of patients with mCRPC in correlation with measures of outcome (ie clinical benefit, Prostate-Specific Androgen (PSA) decline, radiographic response, time to treatment discontinuation), in an effort to identify predictors of response or resistance to therapy.

SECONDARY OUTCOMES:
Eastern Cooperative Oncology Group (ECOG) performance status | Up to 30 weeks
PSA response | Up to 30 weeks
Radiological progression-free survival according to Prostate Cancer Working Group 2 (PCWG2) | Up to 30 weeks or until Disease Progression
Pain status using a numerical rating scale from 0 to 10. | Up to 30 weeks
Time to best clinical benefit (based on pain, analgesic consumption, and performance status) | Up to 30 weeks
Overall survival | Up to 40 months
Explore the potential association between serum PSA with bone marrow (BM) androgen (testosterone, dehydrotestosterone, androstenedione, cortisol, pregnenolone and progesterone) levels and androgen receptor expression while on Cabazitaxel | Up to 30 weeks
Prospective collection of BM biopsies and aspirates to measure the effect of Cabazitaxel on markers of bone metabolism(N-terminal Androgen Receptor(AR),C-terminal AR,splice variant presence,NKX3.1,AR coactivator expression,CYP17,p53,Aurora kinase,UBE2C) | Up to 30 weeks
Correlation between levels of circulating androgens(testosterone, dehydrotestosterone,androstenedione,cortisol,pregnenolone and progesterone)and those in the bone marrow before and during treatment with Cabazitaxel with measures of efficacy | Up to 30 weeks
Number of participants with Serious and Non-Serious Adverse Events graded according to National Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | Up to 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Efstathiou, MD,Ass. Prof, Study Chair — Unit of Medical Oncology,Department of Clinical Theraputics,General Hospital of Athens "Alexandra"
Locations (6):
- Greece (6):
  - Athens Medical Center, Dept of Medical Oncology, Athens, Maroussi
  - EUROMEDICA General Clinic of Thessaloniki, Thessaloniki, Thessaloniki
  - General Hospital of Athens "Alexandra", Unit of Medical Oncology, Dept of Clinical Therapeutics, Athens
  - Agii Anargiri Cancer Hospital, 3rd Dept of Medical Oncology, Athens
  - Ioannina University Hospital, Dept of Medical Oncology, Ioannina
  - Papageorgiou General Hospital, Dept of Medical Oncology, Thessaloniki